CLINICAL TRIAL: NCT01107938
Title: Efficacy and Safety of Ilaprazole for GERD: A Randomized,Double-Blind, Esomeprazole-Controlled,Phase2,Multicenter Trial in China
Brief Title: Ilaprazole for the Treatment of Gastroesophageal Reflux Disease (GERD) in Chinese Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Haitang Hu, Livzon Pharmaceutical Group Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Livzon-IY-81149R-09; SFDA2004L00137
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2010-04

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — ilaprazole; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 10 mg ilaprazole (Experimental)
  Interventions: Drug: 10 mg ilaprazole
- 15 mg ilaprazole (Experimental)
  Interventions: Drug: 15 mg ilaprazole
- 40 mg esomeprazole (Active Comparator)
  Interventions: Drug: 40 mg esomeprazole

INTERVENTIONS:
Drug: 10 mg ilaprazole — Two 5-mg ilaprazole tablets (Livzon Pharm Group Inc., China) together with one placebo tablet of ilaprazole and one placebo tablet of esomeprazole in a package being taken orally each morning on an empty stomach for 8 weeks
  Arms: 10 mg ilaprazole
Drug: 15 mg ilaprazole — Three 5-mg ilaprazole tablets (Livzon Pharm Group Inc., China) together with one placebo tablet of esomeprazole in a package being taken orally each morning on an empty stomach for 8 weeks
  Arms: 15 mg ilaprazole
Drug: 40 mg esomeprazole — One 40-mg esomeprazole tablet (AstraZeneca, Nexium) together with three 5-mg placebo tablets of ilaprazole in a package being taken orally each morning on an empty stomach for 8 weeks
  Arms: 40 mg esomeprazole

SUMMARY:
This study is designed to evaluate the efficacy and tolerability of ilaprazole relative to that of esomeprazole in healing erosive esophagitis and resolving accompanying symptoms of GERD.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients will be eligible for enrollment if they:

  * are 18-70 years of age,
  * have at least one of the two symptoms, heartburn and reflux,
  * have photographically documented erosive esophagitis confirmed by esophagogastroduodenoscopy(EGD), and graded according to the Los Angeles (LA) Classification (A-D), within 5 days before randomization to treatment. Female patients are required to be nonpregnant, nonlactating, postmenopausal, surgically sterilized, or using a medically acceptable form of birth control, as determined by the investigator. Women of child- bearing potential will receive a pregnancy test.

Exclusion Criteria:

* Patients will be ineligible if they:

  * have cancerous or peptic ulcers, Zollinger-Ellison syndrome, varices of esophagus or fundus of stomach
  * have a known history of gastric acid suppression operation, esophageal operation or peptic operation other than simple closure of perforation,
  * have severe complications, severe other diseases of digestive tract such as Crohn's disease and ulcerative colitis, and severe other systemic diseases,
  * have taken proton pump inhibitors within the 5 days or for more than three consecutive days within the two weeks immediately preceding start of study drug,
  * participated in a clinical trial with an investigational drug or device within the past three months,
  * have hypersensitivity or idiosyncratic reaction to ilaprazole, esomeprazole or any other benzimidazole,
  * have alcoholic intemperance, drug addiction or any other improper habits.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients with healed esophagitis at week 8 | week 8

SECONDARY OUTCOMES:
the proportion of patients healed at week 4 | week 4
resolution of clinical symptoms | week 8

CONTACTS AND LOCATIONS:
Overall Officials: Sanren Lin, MD, Principal Investigator — Peking University Third Hospital; Liya Zhou, MD, Principal Investigator — Peking University Third Hospital

REFERENCES:
- [Derived] Xue Y, Qin X, Zhou L, Lin S, Wang L, Hu H, Xia J. A Randomized, Double-blind, Active-Controlled, Multi-center Study of Ilaprazole in the Treatment of Reflux Esophagitis. Clin Drug Investig. 2016 Dec;36(12):985-992. doi: 10.1007/s40261-016-0446-3. PMID 27605258